CLINICAL TRIAL: NCT06843824
Title: A Graphene Far-infrared Intervention Study of Cognitive Status in Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Psychology, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023YFC3605304-1; 2023YFC3605304 (Other Grant/Funding Number: National Key Research and Development projects)
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Mild Cognitive Impairment (MCI); Subjective Cognitive Decrease (SCD); Alzheimer's Disease(AD); Depression/Anxiety Symptoms
Keywords: Graphene Far Infrared Intervention (GFII); Randomized Controlled Trial (RCT); Older Adults; Subjective Cognitive Decrease (SCD); Mild cognitive impairment (MCI); Alzheimer's Disease(AD)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Graphene far infrared intervention group (Experimental): The intervention group used the Graphene Far Infrared Intervention (GFII), in which a caregiver who had undergone standardized training wore a graphene cap that could heat up to 40°C on the elderly. The cap was worn by the elderly for a fixed period of time each day and removed after approximately 40 minutes. During the time of wearing the cap, the elderly can perform any activity (e.g., reading the newspaper, watching TV) within the length of the power cord in a sitting, lying, standing position, etc.
  Interventions: Device: a custom-made graphene therapy cap
- Wear a normal heatable cap group (Placebo Comparator): The placebo control group used ordinary hats that could be heated to about 40°C and were worn to the head of the elderly by caregivers who had undergone standardized training. The elderly wore the heat generating cap for a fixed period of time each day and removed it after about 40 minutes. During the period of wearing the cap, the elderly can sit, lie down, stand in the position of the length of the power cord, and carry out any activities (e.g., reading newspaper, watching TV)
  Interventions: Device: A regular cap that generates heat

INTERVENTIONS:
Device: a custom-made graphene therapy cap — The GFII involved the use of a custom-made graphene therapy cap. The cap consisted of 3 parts: the main body of the cap, the thermostat and the power adapter. One end of the thermostat was connected to the main body of the cap, and the other end was connected to the power adapter; the adapter was plugged into a 220 V household power outlet. This turned on the cap, and the temperature could be adjusted. The light energy conversion rate of the graphene coating material used in the cap reached 90%, generating a temperature of 40 °C. Five caregivers were responsible for providing care for the elderly individuals. We will provided standardized training on the GFII to their caregivers. Each caregiver was responsible for assisting with the intervention of the elderly individuals that they usually cared for.
  Arms: Graphene far infrared intervention group
Device: A regular cap that generates heat — The rest of the procedure is the same as the GFII group, but the cap used is a regular cap that can heat up to 40°C.
  Arms: Wear a normal heatable cap group

SUMMARY:
This study is a 4-week group controlled trial to explore whether graphene far-infrared intervention can improve the cognitive status of older adults presenting with symptoms of Subjective Cognitive Decline (SCD), Mild Cognitive Impairment (MCI), or Alzheimer's Disease (AD), and is dedicated to enhancing the cognitive status of older adults and improving their mental health. Participants were older adults who presented with cognitive problems. Participants were divided into SCD and MCI/AD groups based on their cognitive level, and each group was further divided into a graphene far-infrared intervention group and a placebo control group. We also measured the depression and anxiety levels of the older adults and incidentally observed whether the graphene far-infrared intervention could have a positive impact on their mental health outcomes, which was not the focus of our study.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years and above (age limit may be relaxed to not less than 45 years if there is a special desire to participate in the intervention)
* No barriers to daily communication
* Individuals participating voluntarily

Exclusion Criteria:

* Good cognitive functioning (SCD score of 0)
* Subjective desire to withdraw
* Individuals who reported discomfort opting out during the experimental procedure

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
SCD | Pre-intervention, 2 weeks after the start of the intervention, 4 weeks after the start of the intervention (at which point the intervention ended), 2 weeks after the end of the intervention, and 4 weeks after the end of the intervention (a total of 5 mea
  Depression was assessed by the Self-Rating Scale for Subjective Cognitive Decrease (SCD). The scale consists of 10 items that are scored from 1 (no change) to 3 (significant increase) based on the patient's self-reported subjective cognitive decompensation. A higher total score indicates more severe subjective cognitive decompensation.
MCI/AD | Pre-intervention, 2 weeks after the start of the intervention, 4 weeks after the start of the intervention (at which point the intervention ended), 2 weeks after the end of the intervention, and 4 weeks after the end of the intervention (a total of 5 mea
  Cognitive function was assessed with the short form of the Montreal Cognitive Assessment (s-MoCA). The items are used to examine function in 6 cognitive domains (i.e., visuospatial/executive function, attention, language, abstraction, delayed memory, and orientation). If the number of years of education is less than or equal to 12, the total score is increased by 1 point. The total score ranges from 0 to 18: scores less than or equal to 11 indicate probable mild cognitive impairment (MCI), and scores less than or equal to 4 indicate probable Alzheimer's disease (AD).

SECONDARY OUTCOMES:
depression | Pre-intervention, 2 weeks after the start of the intervention, 4 weeks after the start of the intervention (at which point the intervention ended), 2 weeks after the end of the intervention, and 4 weeks after the end of the intervention (a total of 5 mea
  Depression was assessed with the Patient Health Questionnaire (PHQ-9). The PHQ-9 contains nine items scored on a scale from 0 (not at all) to 3 (almost every day) based on the self-reported frequency of depressive symptoms in the past 2 weeks. The total score ranges from 0 to 27, and scores above 10 indicate probable depression symptoms.
Anxiety | Pre-intervention, 2 weeks after the start of the intervention, 4 weeks after the start of the intervention (at which point the intervention ended), 2 weeks after the end of the intervention, and 4 weeks after the end of the intervention (a total of 5 mea
  Anxiety was assessed with the Chinese version of the Generalized Anxiety Disorder Scale (GAD-7). The 7 items are rated on a 4-point scale ranging from 0 (never) to 3 (almost every day) to assess the frequency of anxiety symptoms in the past 2 weeks. The total score ranges from 0 to 21, and according to the established criteria, scores above 10 indicate probable anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychology, Chinese Academy of Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No